CLINICAL TRIAL: NCT07040137
Title: Phase III Confirmatory Study 3 of KPS-0373 in Patients With Spinocerebellar Degeneration
Brief Title: Confirmatory Study 3 of KPS-0373 in Patients With Spinocerebellar Degeneration
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kissei Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPS1306; jRCT (Registry Identifier: jRCT)
Record Dates: First submitted 2025-06-25; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Spinocerebellar Degeneration
MeSH Terms: conditions — Spinocerebellar Degenerations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KPS-0373 group (Experimental): * Screening period: One placebo tablet is orally administrated once daily after breakfast for 4 weeks.
  * Treatment period: One KPS-0373 2.4 mg tablet is orally administered once daily after breakfast in 24 weeks.
  Interventions: Drug: KPS-0373
- Placebo group (Placebo Comparator): * Screening period: One placebo tablet is orally administrated once daily after breakfast for 4 weeks.
  * Treatment period: One placebo tablet is orally administered once daily after breakfast in 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KPS-0373 — Oral administration
  Arms: KPS-0373 group
Drug: Placebo — Oral administration
  Arms: Placebo group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, phase III study to evaluate the efficacy and safety of KPS-0373 given once daily after breakfast in 142 patients with spinocerebellar degeneration . This study consists of the 4-week screening period, 24-week treatment period, and 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Japanese SCD patients with mild to moderate ataxia

Exclusion Criteria:

* Patients with secondary ataxia
* Patients with clinically significant hepatic, renal, or cardiovascular dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in SARA total score at 24 weeks of treatment period | Up to 24 weeks
  The SARA is a scale that assesses cerebellar ataxia. An evaluator observes the subject's ability to perform motor activities across in 8 individual items: ("gait: 0-8 points," "stance: 0-6 points," "sitting: 0-4 points," "speech disturbance: 0-6 points," "finger chase: 0-4 points," "nose-finger test: 0-4 points," "fast alternating hand movements: 0-4 points," and "heel-shin slide: 0-4 points." The total SARA score ranges from 0 (no ataxia) to 40 (severe ataxia).

SECONDARY OUTCOMES:
Change from baseline in SARA total score | Up to 24 weeks
  The SARA is a scale that assesses cerebellar ataxia. An evaluator observes the subject's ability to perform motor activities across in 8 individual items: ("gait: 0-8 points," "stance: 0-6 points," "sitting: 0-4 points," "speech disturbance: 0-6 points," "finger chase: 0-4 points," "nose-finger test: 0-4 points," "fast alternating hand movements: 0-4 points," and "heel-shin slide: 0-4 points." The total SARA score ranges from 0 (no ataxia) to 40 (severe ataxia).
Symptom Maintenance Ratio (Ratio of Improvement and Stability Cases) based on SARA total score | Up to 24 weeks
  Subjects with the change in total SARA score from baseline of ≤ -1 point are defined as improved subjects, subjects with the change in total SARA score of > -1 point and < 1 point as unchanged subjects, and subjects with improvement and subjects with no change are defined as subjects maintaining symptoms.
Change from baseline in SARA individual scores | Up to 24 weeks
  The SARA is a scale that assesses cerebellar ataxia. An evaluator observes the subject's ability to perform motor activities across in 8 individual items: ("gait: 0-8 points," "stance: 0-6 points," "sitting: 0-4 points," "speech disturbance: 0-6 points," "finger chase: 0-4 points," "nose-finger test: 0-4 points," "fast alternating hand movements: 0-4 points," and "heel-shin slide: 0-4 points." The total SARA score ranges from 0 (no ataxia) to 40 (severe ataxia).
Change from baseline in SF-8 | Up to 24 weeks
  SF-8 is a questionnaire that comprehensively measures health-related QOL. Subjects answer questions in the following 8 items on a scale of 5 or 6: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. A higher score indicates better health in that item.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: Yes
* The Individual Patient Data (IPD) are available upon reasonable request and with permission of Kissei Pharmaceutical Co., Ltd.
  * For a data sharing request for IPD, please contact Kissei Pharmaceutical at rinsyousiken@pharm.kissei.co.jp.
Supporting Information: Study Protocol, SAP